CLINICAL TRIAL: NCT06429618
Title: Effect of a Low-carbohydrate Diet on Outcomes According to Phenotype in Juvenile Polycystic Ovary Syndrome
Brief Title: Adolescent Polycystic Ovary Syndrome on a Low-carbohydrate Diet
Acronym: PCOS
Status: Completed | Type: Observational
Sponsor: Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Mujde Can Ibanoglu, Assoc. Prof, Etlik Zubeyde Hanım Women's Health Care, Training and Research Hospital
Other Study IDs: 01/07 22.01.2024
Record Dates: First submitted 2024-05-18; First posted 2024-05-28 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Polycystic Ovary Syndrome; Adolescent Behavior; Diet Habit
Keywords: phenotype; polycystic ovary syndrome; adolescents; low carbonhydrate diet
MeSH Terms: conditions — Polycystic Ovary Syndrome; Adolescent Behavior; Feeding Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Phenotype A: PHENOTYPE A: Hyperandrogenism + Ovulatory Dysfunction + PCOM
  Interventions: Dietary Supplement: Low carbonhydrate diet
- Phenotype B: PHENOTYPE B: HA+OD
  Interventions: Dietary Supplement: Low carbonhydrate diet
- Phenotype C: PHENOTYPE C: HA+PCOM
  Interventions: Dietary Supplement: Low carbonhydrate diet
- Phenotype D: PHENOTYPE D: OD+PCOM
  Interventions: Dietary Supplement: Low carbonhydrate diet

INTERVENTIONS:
Dietary Supplement: Low carbonhydrate diet — Each patient will receive a 3-month low-carbohydrate (40% CHO) diet from the same dietitian. Whether the patients adhere to the diet and which components the prescribed diet consists of is recorded in detail. After 3 months of standard application, the patient is examined again by the gynecologist and obstetrician at the PCOS clinic.
  Other Names: 0.; 3.month

SUMMARY:
The aim of the study was to investigate the changes in the clinical and biochemical parameters of adolescents on a low-carbohydrate diet in relation to their PCOS phenotype in the 3rd trimester.

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is an endocrine-metabolic disorder characterized by menstrual irregularities, anovulation, clinical and/or biochemical symptoms of hyperandrogenism (hirsutism and/or acne), micropolycystic ovaries, and metabolic abnormalities. In addition, some clinical and laboratory phenotypic features have been defined that were not previously included in the PCOS definition criteria, but which complement the clinical picture and influence the severity and morbidity of the clinical picture. Phenotype A: HA + OD + PCOM; phenotype B: HA + OD; phenotype C: HA + PCOM and phenotype D: OD + PCOM.For adult patients, internationally recognized diagnostic criteria have been developed based on combinations of otherwise unexplained hyperandrogenism, anovulation and polycystic ovary and are covered by the Rotterdam Consensus Criteria. However, in the adolescent age group, the frequency of anovulatory cycles and associated menstrual irregularities, the frequent symptoms of hyperandrogenism and acne vulgaris in the developmental phase, the problems with testosterone measurement and the prevalence of polycystic ovarian morphology in normal adolescents complicate the diagnosis.

PCOS is a serious clinical and psychological problem for adolescent girls. Key interventions include lifestyle modification, including diet, physical activity and weight loss. These measures have been shown to alter the course of the disease in overweight and obese girls. In particular, it is known that high glycemic index carbohydrate intake and glycemic load lead to a rapid rise in blood glucose levels and increased insulin production.

It is therefore thought that reducing the amount of insulin could have a more positive effect on PCOS than the usual carbohydrates. A low-carbohydrate diet is an effective, weight-independent approach in the treatment of metabolic disorders in PCOS patients. With this in mind, this study aimed to evaluate the clinical and biochemical outcomes at month 3 after application of the low-carbohydrate diet in adolescents according to their PCOS phenotype.

ELIGIBILITY:
Inclusion Criteria:

* at least 1 year has passed since menarche
* under 24 years old
* patients who have not received an oral contraceptive method and have given verbal and written informed consent will be included.

Exclusion Criteria:

* over 24 years old
* hyperprolactinemia, Cushing's syndrome, congenital adrenal hyperplasia, thyroid diseases
* neuromuscular, liver, pancreatic or gastrointestinal diseases
* hormonal medication such as antiandrogens, antidiabetics, glucocorticoids, insulin sensitizers or lipid regulators

Ages: 12 Years to 24 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study will be conducted based on the 2018 ESHRE/ASRM guideline:
  1. Oligo and/or anovulation*
  2. Clinical and/or biochemical hyperandrogenism *Oligo and/or anovulation are defined as follows:
     * It is considered normal in the first year after menarche as part of the pubertal transition
     * Between 1-3 years after menarche: < 21 or > 45 days
     * 3 years after menarche - perimenopause: < 21 or > 35 days or < 8 cycles per year
     * 1 year after menarche: >90 days for each menstrual cycle
     * Absence of menstruation at the age of 15 years or 3 years after menarche.
  Identification of phenotype groups:
  PHENOTYPE A: HA+ OD + PCOM PHENOTYPE B: HA+OD PHENOTYPE C: HA+PCOM PHENOTYPE D: OD+PCOM.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2024-09-30 (Actual); Primary Completion 2024-10-07 (Actual); Study Completion 2025-02-25 (Actual)

PRIMARY OUTCOMES:
demographic datas on the study | 3 months
  Age
Evaluation of demographic data | 3 months
  Smoking
Demographic data at month 3 after application of a low-carbohydrate diet according to PCOS phenotypes in adolescents. | 3 months
  Body mass index Calculation of BMI: Height and body weight of the patients were measured using professionally calibrated devices. BMI was calculated using the formula BMI = weight (kg)/height (m)2.
Evaluation of clinical results at month 3 after application of a low-carbohydrate diet according to PCOS phenotypes in adolescents. | 3 months
  waist circumference(centimeters)
Evaluation of degree of hirsutism at month 3 after application of a low-carbohydrate diet according to PCOS phenotypes in adolescents. | 3 months
  degree of hirsutism (Ferriman-Gallwey Hirsutism Scoring Scale; lowest 8 highest: 24)
Hormone results at month 3 after application of a low-carbohydrate diet according to PCOS phenotypes in adolescents. | 3 months
  prolactin (ng/mL)
androstenedione at month 3 after application of a low-carbohydrate diet according to PCOS phenotypes in adolescents. | 3 months
  androstenedione (mosm/kg)
dehydroepiandrosterone sulfate at month 3 after application of a low-carbohydrate diet according to PCOS phenotypes in adolescents. | 3 months
  dehydroepiandrosterone sulfate (DHEA-S) (μg/dL)
TSH at month 3 after application of a low-carbohydrate diet according to PCOS phenotypes in adolescents. | 3 months
  thyroid stimulating hormone (TSH) (mIU/mL)
SHBG at month 3 after application of a low-carbohydrate diet according to PCOS phenotypes in adolescents. | 3 months
  Hormone test results : sex hormone-binding globulin (SHBG)
17-OH progesterone at month 3 after application of a low-carbohydrate diet according to PCOS phenotypes in adolescents. | 3 months
  17-OH progesterone (mIU/mL)
Testosterone at month 3 after application of a low-carbohydrate diet according to PCOS phenotypes in adolescents. | 3 months
  free and total testosterone (ng/mL)
Lipid profile at month 3 after application of a low-carbohydrate diet according to PCOS phenotypes in adolescents. | 3 months
  Lipid profile: Total cholesterol (mg/dL), high-density lipoprotein (HDL) cholesterol (mg/dL), low-density lipoprotein (LDL) cholesterol (mg/dL), triglycerides (mg/dL).
Glucose at month 3 after application of a low-carbohydrate diet according to PCOS phenotypes in adolescents. | 3 months
  fasting blood glucose
Evaluation of insulin resistance at month 3 after application of a low-carbohydrate diet according to PCOS phenotypes in adolescents. | 3 months
  Calculation of insulin resistance: A fasting blood glucose level between 100-125 mg/dl was considered as 'impaired fasting glucose'. A Homeostatic Model Assessment Insulin Resistance (HOMA-IR) value of ≥2.5 was defined as insulin resistance. Insulin resistance was calculated using the formula of the homeostatic model. [HOMA-IR= fasting glucose (mg/dl)xfasting insulin (mIU/mL)/405].

CONTACTS AND LOCATIONS:
Overall Officials: Mujde Can Ibanoglu, Principal Investigator — Ankara Etlik Zubeyde Hanım Women's Health Training and Research Hospital, Ankara, Turkey.
Locations (1):
- Etlik Zübeyde Hanım, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Joham AE, Pena AS. Polycystic Ovary Syndrome in Adolescence. Semin Reprod Med. 2022 Mar;40(1-02):e1-e8. doi: 10.1055/s-0042-1757138. Epub 2022 Sep 12. PMID 36096151
- [Result] Bozdag G, Mumusoglu S, Zengin D, Karabulut E, Yildiz BO. The prevalence and phenotypic features of polycystic ovary syndrome: a systematic review and meta-analysis. Hum Reprod. 2016 Dec;31(12):2841-2855. doi: 10.1093/humrep/dew218. Epub 2016 Sep 22. PMID 27664216